CLINICAL TRIAL: NCT02224937
Title: MELATOX: Evaluation of Percutaneous Dissolvement of Melatonin When Used as Sunscreen; a Randomized, Placebo Controlled, Double-blind Crossover Study on Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Cecilie Scheuer, ph.d.student, Zealand University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2013-003023-10; 2013-003023-10 (EudraCT Number)
Record Dates: First submitted 2014-08-20; First posted 2014-08-25 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Solar Skin Damage
Keywords: Melatonin; Cognitive parameters; pharmacodynamic; pharmacokinetics
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin:Melatonincreme 12,5% (Experimental): Application of melatonincream 12,5% on 80% of the body-surface at start of investigation.
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Application of placebo cream on 80% of the body-surface at start of investigation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin
  Arms: Melatonin:Melatonincreme 12,5%
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the percutaneous transportation and pharmacokinetics of melatonincream 12,5% when used on 80% of the body area. A test battery consisting of blood, saliva, urine samples at 1,2,3,4,5,6,7,8,12,24 and 36 hours after cream application. Cognitive parameters are investigated using KSS, FTT and CRT tests at above mentioned time points.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes
* Age 18-65 years
* No shiftwork
* No intake of caffeine or alcohol one day before investigation, and under the experiment.
* Pittsburgh sleep quality index <5
* Height 165-190 cm
* Weight 53-85 kg

Exclusion Criteria:

* Pregnancy
* Active skin-disease
* Use of hypnotic or sedative drugs.
* Known sleeping disorder
* Known allergy to contents of the cream.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Changes in Karolinska Sleepiness Scale after application of melatonincream 12,5% on 80% of the body-surface area. | 1,2,3,4,5,6,7,8,12,24 and 36 hours post exposure.
  Karolinska sleepiness scale is a valid scale for measurement of subjective sleepiness in individuals.
  This scale is used to detect any changes in subjective sleepiness over a time period of 36 hours after application of melatonincream 12,5% on 80% of the body-surface area.

SECONDARY OUTCOMES:
Changes in continuous reaction time over a time period of 36 hours after application of melatonin cream 12,5% on 80% of the body surface area. | 1,2,3,4,5,6,7,8,12,24 and 36 hours post exposure.
  Continuous reaction time is a neuropsychological test designed to investigate endurance and attention by testing the persons ability to react to external stimuli over a given time period.
  This parameter is used to detect changes in endurance and attention over a time period of 36 hours after application of melatonincream 12,5% on 80% of the body-surface area.
Changes in finger tapping test over a time period of 36 hours after application of melatonin cream 12,5% on 80% of the body surface area. | 1,2,3,4,5,6,7,8,12,24 and 36 hours post exposure.
  Finger tapping test is a simple way to investigate psychomotoric speed and control. Impaired psychomotoric speed is accepted as a predictor for cerebral dysfunction.
  This parameter is used to detect changes in psychomotoric speed and control over a time period of 36 hours after application of melatonincream 12,5% on 80% of the body surface area.
Changes in serum melatonin concentration | 1,2,3,4,5,6,7,8,12,24 and 36 hours post exposure.
  Blood samples are collected at the above mentioned time points. Serum melatonin is evaluated by laboratory tests.
  Blood samples are used to detect the changes in serum melatonin concentration after application of melatonin cream 12,5% on 80% of the body surface area.
Changes in saliva melatonin concentration. | 1,2,3,4,5,6,7,8,12,24 and 36 hours post exposure
  Saliva samples are collected at above mentioned time points. The concentration of melatonin in saliva is tested using laboratory analyses.
  Saliva samples are collected to detect changes in saliva melatonin concentration over a time period of 36 hours after application of melatonincream 12,5% on 80% of the body surface area.
Changes in urine melatonin concentration | 0-4,4-8,8-12,12-24 and 24-36.
  Urine is collected in the above mentioned time intervals, and the concentration of melatonin is found by measuring the concentration of the metabolite 6-sulfatoxymelatonin using RIA.
  The urine samples are collected and used to detect changes in 6-sulfatoxymelatonin concentration over a time period of 36 hours after application of melatonincream on 80% of the body surface area.

OTHER OUTCOMES:
Measurement changes in bloodpressure and puls. | 1,2,3,4,5,6,7,8,12,24 and 36 hours post exposure
  Blood pressure and puls was monitored throughout the study.
Holter monitoring | 1-36 hours
  Registration of alterations in heart rate throughout the time period of 0-36 hours will be continuously monitored using af Holter monitor.
Measurement of changes in body-temperature | 1,12,24 and 36 hours post exposure
  Body-temperature was monitored at 1,12,24 and 36 hours after cream application.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Ms Scheuer, ph.d.student, Principal Investigator — Køge Sygehus
Locations (1):
- Herlev Sygehus, Herlev, Herlev, Denmark